CLINICAL TRIAL: NCT06607406
Title: A Randomized Trial of Accelerated Postoperative Radiotherapy for Intermediate- and High-risk Patients With HNSCC (Head and Neck Squamous Cell Carcinoma) Initiating Radiotherapy Greater Than 6 Weeks After Surgery (PORTRush)
Brief Title: Postoperative Radiotherapy for Intermediate- and High-risk Patients With HNSCC Greater Than 6 Weeks After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00119512; ONC-HN-2406 (Other: Atrium Health)
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: Radiotherapy; Accelerated radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional fractionation (5 Fractions) (Active Comparator): 5 fractions per week, daily treatment Monday-Friday; dosage at the discretion of the treating radiation oncologist per standard of care
  Interventions: Radiation: Conventional radiotherapy
- Accelerated fractionation (6 Fractions) (Experimental): 6 fractions per week, daily treatment plus twice daily treatment for 1 day Monday-Friday; dosage at the discretion of the treating radiation oncologist per standard of care
  Interventions: Radiation: Accelerated radiotherapy

INTERVENTIONS:
Radiation: Accelerated radiotherapy — 6 fractions per week, BID fractions one day per week
  Arms: Accelerated fractionation (6 Fractions)
Radiation: Conventional radiotherapy — 5 fractions per week, daily M-F
  Arms: Conventional fractionation (5 Fractions)

SUMMARY:
The goal of this clinical trial is to determine whether accelerated radiotherapy (involving 6 treatments per week) is better than standard radiotherapy (involving 5 treatments per week) at treating cancer of the head and neck when initiated more than 6 weeks after surgery.

DETAILED DESCRIPTION:
This study is a randomized trial designed to determine the effect of Accelerated Fractionation (AF) versus Conventional Fractionation (CF) PORT on locoregional recurrence-free survival, progression-free survival, overall survival, toxicity, and treatment package time in participants with resected intermediate and high-risk Head and Neck Squamous Cell Carcinoma (HNSCC) planned to start Post Operative Radiotherapy (PORT) greater than six weeks after surgery. Eligible participants in both cohorts will be randomized 1:1 to receive five fractions per week of standard conventional fractionation radiotherapy or six fractions per week of accelerated fractionation radiotherapy. If randomized to the standard conventional fractionation group, participants will be treated with five fractions of radiation per week, received daily. If randomized to the accelerated fractionation group, participants will be treated with 6 fractions of radiotherapy per week, received daily and twice daily treatments on one day of the week.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed head and neck squamous cell carcinoma of the oral cavity, oropharynx, larynx, hypopharynx, sinus, or lymph nodes of the neck of unknown primary.
* Planned for curative intent postoperative radiotherapy based on pathologic risk factors.

  * Patients with non-HPV-mediated oropharyngeal squamous cell carcinoma or non-oropharyngeal squamous cell carcinoma must have at least one of the following: pathologic tumor classification pT3-4, multiple lymph nodes involved with cancer, perineural invasion, lymphovascular invasion, close margins (within 2 mm for oropharyngeal cancer status post transoral resection; within 5 mm for all others) or cleared margins (initially positive, subsequently cleared in an additional specimen), extranodal extension (any extent), or positive surgical margins.
  * Patients with HPV-mediated oropharyngeal squamous cell carcinoma must have at least one of the following pathologic risk factors: extranodal extension (any extent), positive surgical margins, or more than 4 lymph nodes involved with cancer.
* Complete macroscopic surgical resection with curative intent for HNSCC with an anticipated interval between the primary surgical resection and initiation of postoperative radiotherapy greater than 42 days but less than or equal to 112 days from surgery. Note: the start date of the time to initiation of PORT is the first (primary) surgical resection. This does not include diagnostic procedures (e.g., biopsy, diagnostic tonsillectomy) or any subsequent surgical interventions for any reason (e.g., wound complications).
* Age ≥ 18 years at the time of enrollment.
* ECOG performance status of 0-1.
* Ability to understand and the willingness to sign an IRB-approved informed consent document directly, in English or Spanish, and to complete study-related forms and activities.

Exclusion Criteria:

* Recurrent head and neck cancer that has recurred after prior courses of definitive RT or surgery followed by postoperative RT/CRT. Note that individuals who have been treated with surgery alone and are now recurrent are eligible.
* Second primary head and neck cancer after initial treatment of a prior head and neck cancer.
* History of prior radiotherapy to the head and neck region, such that any portion of the anticipated target volume overlaps with any region that was previously targeted.
* Active malignancy other than the head and neck cancer to be treated with PORT (excluding non-melanoma skin cancer, in situ carcinoma of any site).
* Metastatic disease from the head and neck cancer to be treated with PORT defined as distant organ involvement outside of the head and neck and/or non-regional lymph node involvement outside of the head and neck.
* Time from primary surgical resection to anticipated initiation of PORT greater than 112 days.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Not a candidate for radiation therapy per treating clinician. For example, individuals who are pregnant or plan to become pregnant (due to the risks of the developing fetus) or any other contraindication to radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional Recurrence-free Survival | 2 years post radiotherapy
  Time to locoregional recurrence, will be assessed on an intention to treat basis using a one-sided log rank test to compare hazard rates between groups. Kaplan-Meier survival curves will also be generated with locoregional failure or death as the event of interest and last clinical disease assessment as a right-censor.

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 5 years
  Progression-free survival will be calculated from the time of randomization to disease recurrence or death from any cause as the event and last follow-up as a right-censor. It will be compared between treatment arms.
Overall survival (OS) | up to 5 years
  Overall survival will be calculated from the time of randomization to death from any cause, with last follow-up as a right-censor.
Acute and late toxicities | up to 24 months post radiotherapy
  Acute and late toxicities between each treatment arm will be measured by evaluating adverse events (AEs) by grade in each treatment arm. Using the Chi-square test (or Fisher's exact test if cell frequencies <5) and a significance level of 0.05, comparisons will be made of the following outcomes between treatment arms: 1) the number of participants with at least one AE of grade 3 or higher, 2) the number of participants with grade 1 or higher toxicity, and 3) the number of patients with grade 3 or higher toxicity. Each of these analyses will result in the construction of 2x2 tables thus the use of the Chi-Square (or Fisher's exact test) will be appropriate. These analyses will be completed for both acute (between RT start and 90 days after RT) and late (more than 90 days after RT completion) toxicities.
Patient Report Outcomes (PRO) - PRO-CTCAE | at baseline, end radiotherapy (RT), 3, 6, 12, and 24-months post RT
  PRO-CTCAE measure of toxicity will be assessed by describing the counts and frequencies for the worst score observed in each participant in the whole cohort and by treatment arm. Using the Chi-square test (or Fisher's exact test if cell frequencies <5) and a significance level of 0.05, a comparison will occur of the following outcomes between treatment arms: 1) the number of patients with at least one PRO-CTCAE score of grade 1 or higher, and 2) the number of patients with at least one PRO-CTCAE score of grade 3 or higher. These comparisons 1 and 2 will be completed for both acute (between RT start and 90 days after RT) and late (more than 90 days after RT completion) toxicities. The analysis of change in PRO-CTCAE score over time will also be performed using a likelihood-based Generalized Linear Mixed Model (GLMM) approach.
Patient Reported Outcomes (PRO) - MDASI-HN | at End of Radiotherapy (RT), 3, 6, 12, and 24-months post RT
  The MDASI-HN is a 28-item measure with three subscales: the 13 core MDASI items, 9 head and neck cancer-specific items, and 6 items specific to interference in daily life by the patient's symptoms. The change from baseline at each time point will be summarized using mean and standard deviation at end RT, 3, 6, 12, and 24-months post RT.
Nutritional Toxicity | up to 24 months post Radiotherapy
  Nutritional toxicity will be measured by comparing the rates of reactive gastrostomy tube placement using a Fisher's exact test. For patients in whom a feeding tube is placed, the duration of tube will be defined as the time from tube placement to removal or last follow-up with a tube (right-censor) and will be estimated using the Kaplan-Meier method and compared between groups using the log-rank statistics.
Time to initiation of Postoperative Radiotherapy (PORT) | up to 16 weeks
  Time to initiation of PORT will be calculated as the number of days from date of primary curative resection (surgery date = day 0) to initiation of RT. This value will be compared between groups using a 2-sample t-test to see if there is a significant difference between groups on this covariate.
Treatment package time | from surgical resection to end of PORT - up to approx. 165 days
  The treatment package time will be calculated as the number of days from the primary surgical resection to the end of PORT (the last RT treatment for participants who complete therapy; for participants who do not complete the prescribed course of RT, this metric is moot) and compared between groups using a 2-sample T-test. The proportion of patients with treatment package time less than 100 days will be determined and compared between groups using the Chi-square test (or Fisher's exact test if cell frequencies <5).
Demographic characteristics of eligible participants | Prior to Radiotherapy (Pre-screening and baseline)
  The characteristics (age, gender assigned at birth, race, ethnicity) of potentially eligible participants will be described using count and frequency for categorical variables and mean (standard deviation) and median (range) for continuous variables. These factors will be compared between groups who do and do not enroll on study using the Chi-square tests for categorical and 2-sample t-tests for continuous measures. For participants who choose not to enroll, the reasons and rationale provided to support that decision will be described using count and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hughes, MD, Principal Investigator — Atrium Health Wake Forest Baptist Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Advocate Aurora Radiation Oncology, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No